CLINICAL TRIAL: NCT06385834
Title: The Effect of Morning vs Evening Aerobic Exercise Training on Cardiac Remodeling and Function Improvement in Patients After ST Elevation Myocardial Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jun Pu, professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY2014-041-A
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: Circadian rhythm; ST-segment Elevation Myocardial Infarction; Aerobic exercise
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: The study was divided into three groups: morning intervention group (8:00-9:00AM), evening intervention group (16:00-17:00AM) and control group
Who Masked: Outcomes Assessor
Masking Description: In this study, outcome measurement personnel and intervention personnel were separated during the whole process of the experiment, outcome measurement personnel did not know the grouping status, intervention personnel and rehabilitation therapists did not participate in the outcome measurement work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning rehabilitation group (Experimental): Patients were randomly assigned to the morning rehabilitation group（8:00-9:00AM） for a 12-week outpatient training program that included a combination of warm-up, aerobic, and relaxation exercises three times a week.
  Interventions: Other: Morning aerobic exercise
- Evening rehabilitation group (Experimental): Patients were randomly assigned to an Evening rehabilitation group(16:00-17:00PM) for a 12-week outpatient training program that included a combination of warm-up, aerobic, and relaxation exercises three times a week.
  Interventions: Other: Evening aerobic exercise
- Control group (No Intervention): Patients randomly assigned to the control group will receive standard care, regular follow-up, optimized medication, and recommendations for a healthy lifestyle.

INTERVENTIONS:
Other: Morning aerobic exercise — Patients were randomly assigned to morning aerobic exercise training for a 12-week outpatient training program that included a combination of warm-up, aerobic, and relaxation exercises three times a week. Each class consists of 10 minutes of warm-up training, 40 minutes of aerobic training and 10 minutes of relaxation training. The intensity of aerobic exercise training will be personalized. According to the guidance of relevant guidelines, the exercise intensity of patients will be determined according to the results of their first cardiopulmonary exercise experiment, and the exercise load will be gradually increased according to the exercise program until the predetermined goal is reached. Patient fatigue levels will be monitored throughout the exercise using the borg scale.
  Arms: Morning rehabilitation group
Other: Evening aerobic exercise — Patients were randomly assigned to evening aerobic exercise training for a 12-week outpatient training program that included a combination of warm-up, aerobic, and relaxation exercises three times a week. Each class consists of 10 minutes of warm-up training, 40 minutes of aerobic training and 10 minutes of relaxation training. The intensity of aerobic exercise training will be personalized. According to the guidance of relevant guidelines, the exercise intensity of patients will be determined according to the results of their first cardiopulmonary exercise experiment, and the exercise load will be gradually increased according to the exercise program until the predetermined goal is reached. Patient fatigue levels will be monitored throughout the exercise using the borg scale.
  Arms: Evening rehabilitation group

SUMMARY:
The aim of the study was to intervene in the Aerobic exercise time of patients with STEMI and to explore the optimal exercise time for STEMI patients

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the first cause of mortality worldwide. More than 30% of CVD-connected fatalities are ascribed to ST-segment Elevation myocardial infarction (STEMI). There is strong and consistent evidence that aerobic exercise after a STEMI improves overall and cardiovascular-related mortality. Aerobic exercise (AE) acts in key mechanisms of cardiac remodeling and function improvement after STEMI, thus contributing both to prevent or postpone harmful adaptations, and even to recover from negative alterations caused by cardiac ischemia. However, the time of day to exercise for STEMI patients' optimal cardiac benefits is currently unknown.

The circadian clock endows the host with temporal precision and robust adaptation to the surrounding environment. Almost all physiologic, metabolic and endocrine processes, including glycolysis, lipid and carbohydrate metabolism as well as cardiovascular function (heart rate, blood pressure) are influenced by the circadian clock. Recent investigations in rodents utilizing gain-of-function/loss-of-function models and in humans have identified Adverse cardiovascular events have day/night patterns is related to endogenous circadian clock control of platelet activation events. Several studies have also demonstrated the effect of AE at different times on blood pressure. Indeed, timing is critical in amplifying the beneficial impact of AE. However, these studies did not address cardiac structural remodeling or other CVD-related metabolic markers, it difficult to determine the physiological and structural effects of different time AE on cardiovascular health.

Thus, In this trial our aim is to assess, in patients who have had an STEMI, AE in which time of a day can give the best benefits to cardiac remodeling and function improvement.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75-years-old;
* Typical symptoms of acute myocardial infarction within 24 hours, with ST segment elevation of ≥1mm in two consecutive leads on electrocardiogram
* After receiving complete revascularization treatment
* Cardiac function grading I to II without any other serious complications
* Left ventricular ejection fraction >30%
* Compliant with the guidelines of the American College of Cardiology/American Heart Association for participating in cardiac rehabilitation standards
* Signed written informed consent.

Exclusion Criteria:

* Patients with unstable angina
* severe symptomatic congestive heart failure detectable myocardial ischemia
* valvular disease requiring surgery
* severe ventricular arrhythmias
* severe concomitant life-threatening diseases such as cancer, and rheumatoid disease
* osteoarticular diseases that may affect the exercise process

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
left ventricle ejection fraction | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Use cardiac ultrasound system to measure left ventricle ejection fraction

SECONDARY OUTCOMES:
Oxygen consumption | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Patients will be submitted to cardiopulmonary exercise testing on a bicycle, using the modified Bruce protocol. Expired gases will be continuously collected throughout exercise and analyzed for ventilatory volume (VE) and for oxygen (O2) and carbon dioxide (CO2) content, using dedicated analyzers. The investigators will assess exercise capacity mainly by measuring anaerobic threshold oxygen consumption and peak oxygen consumption.
Endothelial Function | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Use high-resolution Doppler duplex ultrasound e equipment to analysis Baseline arterial diameter (mm), peak arterial diameter (mm).
Skeletal muscle and fat mass | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Determined by multifrequency BIA using an InBody 770 analyzer (InBody Co., Ltd), that estimate skeletal muscle mass, Body fat mass, distribution of lean body mass and ratio of segmental lean mass.
Cardiac structure | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Use cardiac ultrasound system to measure left ventricular end-diastolic/end-systolic internal diameter, and left ventricular anterior wall thickness.
One year major Adverse Cardiovascular Events | From baseline to one year after participating in rehabilitation
  All patients were followed to major adverse cardiovascular events occurred. The investigators observed the incidence of major adverse cardiovascular events during follow-up, including recurrent myocardial infarction, new heart failure, intractable angina and cardiac death.
VE/VCO2-SLOPE | at baseline，at the sixth week, and after the 12th week of training or follow-up
  Patients will be submitted to cardiopulmonary exercise testing on a bicycle, using the modified Bruce protocol. Expired gases will be continuously collected throughout exercise and analyzed for ventilatory volume (VE) and for oxygen (O2) and carbon dioxide (CO2) content, using dedicated analyzers. The VE/VCO2-SLOPE will be collected.
Flow-mediated dilation | at baseline, at the sixth week, and after the 12th week of training or follow-up
  Use high-resolution Doppler duplex ultrasound e equipment to analysis FMD (%)-formula (peak diameter-baseline diameter) / (baseline diameter) *100.
glucose | at baseline, at the sixth week, and after the 12th week of training or follow-up
  A fasting venous blood sample will be obtained immediately before and after the study for measurement of glucose.
Blood lipid | at baseline, at the sixth week, and after the 12th week of training or follow-up
  A fasting venous blood sample will be obtained immediately before and after the study for measurement of total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides.
N-terminal pro-BNP | at baseline, at the sixth week, and after the 12th week of training or follow-up
  A fasting venous blood sample will be obtained immediately before and after the study for measurement of N-terminal pro-BNP.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China